CLINICAL TRIAL: NCT02883855
Title: Impact of Graft Thickness on Visual Gain After Descemet's Stripping Automated Endothelial Keratoplasty
Acronym: EP-GREFF
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Régional Metz-Thionville (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-08Obs-CHRMT
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-09-15 (Estimated); Status verified 2016-08

CONDITIONS: DSAEK Patient

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
The aim of this study to determinate if there is a correlation between visual acuity gain in patients who underwent a Descemet's stripping automated endothelial keratoplasty (DSAEK) corneal keratoplasty and the central thickness of the graft.

DETAILED DESCRIPTION:
Were included in this study eyes who underwent a DSAEK for endothelial dysfunctions indication (mainly acquired after phacoemulsification or for Fuchs dystrophy) between early 2012 and mid 2015 at CHR Metz-Thionville (Mercy Hospital) Were excluded eyes presenting pathologies (e.g. Age-Related Macular Degeneration, or diabetic macular edema) which are known to induce visual acuity decrease, non-related to the success of the graft and graft failure cases. Central graft thickness was measured in Anterior Segment Optical Coherence Topography (AS-OCT RS-3000 Nidek). Visual acuity gain was defined by the differential between pre-operative visual acuity (VA) and post operative best corrected visual acuity (BCVA) obtained during post-operative visits.

ELIGIBILITY:
Inclusion Criteria:

* patients with endothelial dysfunctions indication

Exclusion Criteria:

- eyes presenting pathologies (e.g. Age-Related Macular Degeneration, or diabetic macular edema) which are known to induce visual acuity decrease, non-related to the success of the graft and graft failure cases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Were included in this study eyes who underwent a DSAEK for endothelial dysfunctions indication (mainly acquired after phacoemulsification or for Fuchs dystrophy) between early 2012 and mid 2015 at CHR Metz-Thionville (Mercy Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2015-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Visual acuity gain after DSAEK lamellar keratoplasty | 1 year